CLINICAL TRIAL: NCT01155739
Title: Etude Prospective Sur l'Impact de l'Utilisation de la Procalcitonine Dans l'évaluation de la Poursuite ou de l'arrêt du Traitement Antibiotique Empirique Lors de péritonites et d'Infections Intra-abdominales
Brief Title: Procalcitonin as a Marker for the Length of Antibiotic Treatment in Peritonitis and Intra-abdominal Infections
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, professor of surgery, University of Lausanne Hospitals
Other Study IDs: 141/08, Propéritonite
Record Dates: First submitted 2009-07-23; First posted 2010-07-02 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Secondary or Tertiary Peritonitis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- procalcitonine monitoring: PCT group: antibiotic use is tailored by serum procalcitonin values, determined every 48houres.
- control group: control group: antibiotic use and length of treatment as defined by guidelines

SUMMARY:
Procalcitonin level used for determining length of antibiotic treatment in peritonitis and intra-abdominal infections. Hypothesis is that length of antibiotic use can be shortened by this method.

DETAILED DESCRIPTION:
Prospective randomized trial

ELIGIBILITY:
Inclusion Criteria:

* More than 18 yo
* Patient requiring surgery for peritonitis or intra-abdominal infection following: perforation, necrosis, previous operation...
* Mannheim Peritonitis score > 14
* SIRS present
* Probability of survival > 72h
* Informed consent by patient/relatives

Exclusion Criteria:

* No SIRS
* Long date corticoid treatment
* Immunosuppression
* Thyroid medullary carcinoma
* Anaphylactic shock
* Acute hepatic deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with SIRS due to peritonitis or intra-abdominal infections
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2009-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
antibiotic treatment length, hospitalisation length without antibiotic, infection recurrence, antibiotic cost | at one month and during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Steve Aellen, MD, Principal Investigator — Department of visceral surgery, university hospital
Locations (1):
- University Hospital of Lausanne, Lausanne, Switzerland